CLINICAL TRIAL: NCT01350362
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 4-arm, 26 Week Parallel-Group Study to Evaluate Efficacy, Safety and Tolerability of 2 Oral Doses and 2 Regimes of Tideglusib vs Placebo in Mild-to-Moderate AD Patients
Brief Title: Efficacy, Safety and Tolerability of Tideglusib to Treat Mild-to-Moderate Alzheimer's Disease Patients
Acronym: ARGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noscira SA (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP031112-10B04
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Alzheimer's Disease
Keywords: tideglusib; Alzheimer; NP-12; NP031112; ARGO; Noscira
MeSH Terms: conditions — Alzheimer Disease | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tideglusib 1000 mg Q.D. (Experimental): Group dosed with 1000 mg once daily for 26 weeks/extension
  Interventions: Drug: tideglusib
- Tideglusib 1000 mg Q.O.D. (Experimental): Group dosed with 1000 mg once every other day for 26 weeks/extension
  Interventions: Drug: tideglusib
- Tideglusib 500 mg Q.D. (Experimental): Group dosed with 500 mg once daily for 26 weeks/extension
  Interventions: Drug: tideglusib
- Placebo (Placebo Comparator): Once daily administration for 26 weeks/extension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tideglusib — 1000 mg of tideglusib as a powder for oral suspension once daily in an overnight fasted state for 26 weeks/extension.
  Other Names: NP-12; NP031112
  Arms: Tideglusib 1000 mg Q.D.
Drug: tideglusib — 1000 mg of tideglusib as a powder for oral suspension once every other day in an overnight fasted state for 26 weeks/extension
  Other Names: NP-12; NP031112
  Arms: Tideglusib 1000 mg Q.O.D.
Drug: tideglusib — 500 mg of tideglusib as a powder for oral suspension once daily in an overnight fasted state for 26 weeks/extension.
  Other Names: NP-12; NP031112
  Arms: Tideglusib 500 mg Q.D.
Drug: Placebo — Powder for oral suspension administered once daily in an overnight fasted state for 26 weeks/extension.
  Other Names: NP-12; NP031112
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the cognitive changes after administration of tideglusib versus placebo at two oral doses and two treatment regimes for 26 weeks in patients with mild to moderate Alzheimer's disease.

After the 26 week core treatment period, the patients may continue in the study under blinded conditions for an optional extension period up to a maximum of 39 additional weeks (total study duration up to 65 weeks), until the last patient in the study has completed the 26 week of treatment.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled, randomized, parallel group study will be conducted at multiple centers in the European Union. Patients with mild to moderate Alzheimer's disease will undergo a screening period, and then they will be randomized to one of these four groups: tideglusib 1000 mg once daily (Q.D.), tideglusib 1000 mg every other day (Q.O.D.), tideglusib 500 mg Q.D., or matching placebo, for a 26-week, double-blind, placebo-controlled treatment period.

ELIGIBILITY:
Main Inclusion Criteria:

1. Men and women (of non-childbearing potential) with a diagnosis of probable Alzheimer's disease.
2. Age of 50 to 85 years.
3. MMSE score 14 to 26.
4. Well-tolerated treatment with one of the approved Acetylcholinesterase-Inhibitors and/or Memantine in a stable dose

Main Exclusion Criteria:

1. Significant psychiatric on medical disease.
2. Any chronic liver disease as indicated by out of range values of ALAT, ASAT or direct bilirubin, clinically relevant hepatic steatosis or other clinical manifestations of liver disease
3. Chronic daily drug intake of excluded concomitant medications.
4. Enrollment in another investigational drug study within 3 months before the baseline visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog+ | 26 weeks
  The change from Baseline of the 3 active study medication groups will be compared with the placebo group in Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog+)

SECONDARY OUTCOMES:
Adverse events (AEs): Number of AEs and patients with an incidence rate of ≥ 5% AEs | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Alzheimer's Disease Cooperative Study Unit Activities of Daily Living (ADCS-ADL). | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Mini Mental State Examination (MMSE) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Word Fluency test | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Neuropsychiatric Inventory (NPI) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Geriatric Depression Scale (GDS) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Clinical Global Impression of Change (CGIC) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the European Quality of life Instrument (EQ-5D) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Caregiver time (RUD Lite) | 26 weeks
Change from Baseline of the 3 active study medication groups will be compared with the placebo group in the Questionnaire on urinary incontinence | 26 weeks
Exploratory Endpoints (only in a subgroup of patients at predefined sites): Change from Baseline of the 3 active study medication groups will be compared with the placebo group in levels of τ, phospho-τ, and β-amyloid in CSF and change in MRI measures. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teodoro del Ser, PhD, Study Director — Noscira SA
Locations (6):
- Leuven and 4 Additional Cities, Belgium
- Turku and 3 Additional Cities, Finland
- Paris and 10 Additional Cities, France
- Freiburg and 5 Additional Cities, Germany
- Madrid and 7 Additional Cities, Spain
- London and 11 Additional Cities, United Kingdom